CLINICAL TRIAL: NCT04640038
Title: Contrast Enhanced Ultrasound (CEUS) Detection of Microvascular Perfusion Impairment in COVID-19 Pediatric Patients
Brief Title: Contrast Enhanced Ultrasound in COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Misun Hwang, MD, Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-017501
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Covid19; Multisystem Inflammatory Syndrome in Children (MIS-C)
Keywords: Ultrasound; Contrast-enhanced ultrasound
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Contrast-enhanced Ultrasonography (Experimental): Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection (if there are two injections of contrast) of the contrast agent.
  Interventions: Drug: Sulfur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride lipid-type A microspheres — Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed to evaluate for dynamic bowel perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.

SUMMARY:
Initial data from COVID-19 patients suggests that one of the primary causes of death is significant endothelial injury leading to blood clotting and impaired multiorgan microvascular perfusion. The current study uses a safe, convenient bedside imaging tool called contrast-enhanced ultrasound (CEUS) to estimate the extent of microvascular perfusion impairment in the heart, kidneys and/or brain of COVID-19 pediatric patients in vivo and assess the significance of imaging findings by correlating to clinical outcomes.

This pilot study will be conducted at one site, The Children's Hospital of Philadelphia. The investigators plan to enroll and evaluate 30 patients.

DETAILED DESCRIPTION:
The current study uses a safe, convenient bedside imaging tool called contrast-enhanced ultrasound (CEUS) to measure the extent of microvascular perfusion impairment in the heart, kidneys and/or brain of COVID-19 pediatric patients and, as exploratory analysis, to assess the significance of imaging findings by correlating to clinical outcomes.

Sulfur hexafluoride lipid-type A microspheres (LumasonTM, Bracco Inc) is an FDA-approved ultrasound contrast agent. Contrast-enhanced ultrasound scan with a duration of approximately 15 minutes will be performed when a COVID-19 diagnosis has been made (or is highly suspected) according to established clinical procedures. One CEUS will be performed per patient, with up to 2 intravenous injections of the contrast agent. The dosing plan will be weight-adjusted, based on a dose of 0.03 mL/kg (with a maximum dose of 2.4 mL per injection). Organ perfusion will be evaluated in the heart, kidneys, and/or brain. Clinical outcomes during hospital stay will be collected for correlation to CEUS-based measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male/female) hospitalized at the Children's Hospital of Philadelphia (CHOP).
2. Patient 17 years of age or younger.
3. Diagnosis of COVID-19 or high clinical suspicion for COVID-19 despite negative tests (according to the definition of probable case by the European Centre for Disease Prevention and Control).
4. Patients have evidence of cardiovascular compromise, myocardial injury, acute kidney injury and/or new-onset neurological symptoms.
5. Parental/guardian permission (informed consent)

Exclusion Criteria:

1. Medical history of Lumason hypersensitivity

Ages: 1 Minute to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belhadjer Z, Meot M, Bajolle F, Khraiche D, Legendre A, Abakka S, Auriau J, Grimaud M, Oualha M, Beghetti M, Wacker J, Ovaert C, Hascoet S, Selegny M, Malekzadeh-Milani S, Maltret A, Bosser G, Giroux N, Bonnemains L, Bordet J, Di Filippo S, Mauran P, Falcon-Eicher S, Thambo JB, Lefort B, Moceri P, Houyel L, Renolleau S, Bonnet D. Acute Heart Failure in Multisystem Inflammatory Syndrome in Children in the Context of Global SARS-CoV-2 Pandemic. Circulation. 2020 Aug 4;142(5):429-436. doi: 10.1161/CIRCULATIONAHA.120.048360. Epub 2020 May 17. PMID 32418446
- [Background] Abdel-Mannan O, Eyre M, Lobel U, Bamford A, Eltze C, Hameed B, Hemingway C, Hacohen Y. Neurologic and Radiographic Findings Associated With COVID-19 Infection in Children. JAMA Neurol. 2020 Nov 1;77(11):1440-1445. doi: 10.1001/jamaneurol.2020.2687. PMID 32609336
- [Background] Ellul MA, Benjamin L, Singh B, Lant S, Michael BD, Easton A, Kneen R, Defres S, Sejvar J, Solomon T. Neurological associations of COVID-19. Lancet Neurol. 2020 Sep;19(9):767-783. doi: 10.1016/S1474-4422(20)30221-0. Epub 2020 Jul 2. PMID 32622375
- [Background] Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 31;368:m1295. doi: 10.1136/bmj.m1295. No abstract available. PMID 32234718
- [Background] Chen L, Li X, Chen M, Feng Y, Xiong C. The ACE2 expression in human heart indicates new potential mechanism of heart injury among patients infected with SARS-CoV-2. Cardiovasc Res. 2020 May 1;116(6):1097-1100. doi: 10.1093/cvr/cvaa078. Erratum In: Cardiovasc Res. 2020 Oct 1;116(12):1994. doi: 10.1093/cvr/cvaa157. PMID 32227090
- [Background] Yao XH, Li TY, He ZC, Ping YF, Liu HW, Yu SC, Mou HM, Wang LH, Zhang HR, Fu WJ, Luo T, Liu F, Guo QN, Chen C, Xiao HL, Guo HT, Lin S, Xiang DF, Shi Y, Pan GQ, Li QR, Huang X, Cui Y, Liu XZ, Tang W, Pan PF, Huang XQ, Ding YQ, Bian XW. [A pathological report of three COVID-19 cases by minimal invasive autopsies]. Zhonghua Bing Li Xue Za Zhi. 2020 May 8;49(5):411-417. doi: 10.3760/cma.j.cn112151-20200312-00193. Chinese. PMID 32172546
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Wan Y, Shang J, Graham R, Baric RS, Li F. Receptor Recognition by the Novel Coronavirus from Wuhan: an Analysis Based on Decade-Long Structural Studies of SARS Coronavirus. J Virol. 2020 Mar 17;94(7):e00127-20. doi: 10.1128/JVI.00127-20. Print 2020 Mar 17. PMID 31996437
- [Background] Cheng Y, Luo R, Wang K, Zhang M, Wang Z, Dong L, Li J, Yao Y, Ge S, Xu G. Kidney disease is associated with in-hospital death of patients with COVID-19. Kidney Int. 2020 May;97(5):829-838. doi: 10.1016/j.kint.2020.03.005. Epub 2020 Mar 20. PMID 32247631
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Dolhnikoff M, Duarte-Neto AN, de Almeida Monteiro RA, da Silva LFF, de Oliveira EP, Saldiva PHN, Mauad T, Negri EM. Pathological evidence of pulmonary thrombotic phenomena in severe COVID-19. J Thromb Haemost. 2020 Jun;18(6):1517-1519. doi: 10.1111/jth.14844. No abstract available. PMID 32294295
- [Background] Magro C, Mulvey JJ, Berlin D, Nuovo G, Salvatore S, Harp J, Baxter-Stoltzfus A, Laurence J. Complement associated microvascular injury and thrombosis in the pathogenesis of severe COVID-19 infection: A report of five cases. Transl Res. 2020 Jun;220:1-13. doi: 10.1016/j.trsl.2020.04.007. Epub 2020 Apr 15. PMID 32299776
- [Background] Fox SE, Akmatbekov A, Harbert JL, Li G, Quincy Brown J, Vander Heide RS. Pulmonary and cardiac pathology in African American patients with COVID-19: an autopsy series from New Orleans. Lancet Respir Med. 2020 Jul;8(7):681-686. doi: 10.1016/S2213-2600(20)30243-5. Epub 2020 May 27. PMID 32473124
- [Background] GOLD E, CARVER DH, HEINEBERG H, ADELSON L, ROBBINS FC. Viral infection. A possible cause of sudden, unexpected death in infants. N Engl J Med. 1961 Jan 12;264:53-60. doi: 10.1056/NEJM196101122640201. No abstract available. PMID 13706404
- [Background] Ma F, Cang Y, Zhao B, Liu Y, Wang C, Liu B, Wu T, Song Y, Peng A. Contrast-enhanced ultrasound with SonoVue could accurately assess the renal microvascular perfusion in diabetic kidney damage. Nephrol Dial Transplant. 2012 Jul;27(7):2891-8. doi: 10.1093/ndt/gfr789. Epub 2012 Apr 24. PMID 22532616
- [Background] Cao W, Cui S, Yang L, Wu C, Liu J, Yang F, Liu Y, Bin J, Hou FF. Contrast-Enhanced Ultrasound for Assessing Renal Perfusion Impairment and Predicting Acute Kidney Injury to Chronic Kidney Disease Progression. Antioxid Redox Signal. 2017 Dec 10;27(17):1397-1411. doi: 10.1089/ars.2017.7006. Epub 2017 Aug 22. PMID 28715949
- [Background] Putz FJ, Erlmeier A, Wiesinger I, Verloh N, Stroszczynski C, Banas B, Jung EM. Contrast-enhanced ultrasound (CEUS) in renal imaging at an interdisciplinary ultrasound centre: Possibilities of dynamic microvascularisation and perfusion. Clin Hemorheol Microcirc. 2017;66(4):293-302. doi: 10.3233/CH-179103. PMID 28527200
- [Background] Schneider AG, Goodwin MD, Schelleman A, Bailey M, Johnson L, Bellomo R. Contrast-enhanced ultrasound to evaluate changes in renal cortical perfusion around cardiac surgery: a pilot study. Crit Care. 2013 Jul 12;17(4):R138. doi: 10.1186/cc12817. PMID 23849270
- [Background] Goyal A, Yu FTH, Tenwalde MG, Chen X, Althouse A, Villanueva FS, Pacella JJ. Inertial Cavitation Ultrasound with Microbubbles Improves Reperfusion Efficacy When Combined with Tissue Plasminogen Activator in an In Vitro Model of Microvascular Obstruction. Ultrasound Med Biol. 2017 Jul;43(7):1391-1400. doi: 10.1016/j.ultrasmedbio.2017.02.013. Epub 2017 Apr 7. PMID 28395964
- [Background] Istvanic F, Yu GZ, Yu FTH, Powers J, Chen X, Pacella JJ. Sonoreperfusion therapy for microvascular obstruction: A step toward clinical translation. Ultrasound Med Biol. 2020 Mar;46(3):712-720. doi: 10.1016/j.ultrasmedbio.2019.11.011. Epub 2020 Jan 7. PMID 31924423
- [Background] Hwang M. Introduction to contrast-enhanced ultrasound of the brain in neonates and infants: current understanding and future potential. Pediatr Radiol. 2019 Feb;49(2):254-262. doi: 10.1007/s00247-018-4270-1. Epub 2018 Oct 23. PMID 30353273
- [Background] Hwang M, Riggs BJ, Katz J, Seyfert D, Northington F, Shenandoah R, Burd I, McArthur J, Darge K, Thimm MA, Huisman TAGM. Advanced Pediatric Neurosonography Techniques: Contrast-Enhanced Ultrasonography, Elastography, and Beyond. J Neuroimaging. 2018 Mar;28(2):150-157. doi: 10.1111/jon.12492. Epub 2017 Dec 27. PMID 29280236
- [Background] Hwang M, De Jong RM Jr, Herman S, Boss R, Riggs B, Tekes-Brady A, Spevak M, Poretti A, Soares BP, Bailey CR, Dunn E, Shin SS, Shrot S, Huisman TAGM. Novel Contrast-Enhanced Ultrasound Evaluation in Neonatal Hypoxic Ischemic Injury: Clinical Application and Future Directions. J Ultrasound Med. 2017 Nov;36(11):2379-2386. doi: 10.1002/jum.14289. Epub 2017 Jun 26. PMID 28649730
- [Background] Hwang M, Riggs BJ, Saade-Lemus S, Huisman TA. Bedside contrast-enhanced ultrasound diagnosing cessation of cerebral circulation in a neonate: A novel bedside diagnostic tool. Neuroradiol J. 2018 Dec;31(6):578-580. doi: 10.1177/1971400918795866. Epub 2018 Sep 7. PMID 30189812
- [Background] Hwang M, Sridharan A, Darge K, Riggs B, Sehgal C, Flibotte J, Huisman TAGM. Novel Quantitative Contrast-Enhanced Ultrasound Detection of Hypoxic Ischemic Injury in Neonates and Infants: Pilot Study 1. J Ultrasound Med. 2019 Aug;38(8):2025-2038. doi: 10.1002/jum.14892. Epub 2018 Dec 17. PMID 30560547
- [Background] Benjamin JL, Dennis R, White S Jr, Munson D, Anupindi SA, Piskunowicz M, Darge K, Gokli A, Hwang M. Improved Diagnostic Sensitivity of Bowel Disease of Prematurity on Contrast-Enhanced Ultrasound. J Ultrasound Med. 2020 May;39(5):1031-1036. doi: 10.1002/jum.15168. Epub 2019 Nov 9. PMID 31705672
- [Background] Hwang M, Hariri G, Lyshchik A, Hallahan DE, Fleischer AC. Correlation of quantified contrast-enhanced sonography with in vivo tumor response. J Ultrasound Med. 2010 Apr;29(4):597-607. doi: 10.7863/jum.2010.29.4.597. PMID 20375378
- [Result] Tierradentro-Garcia LO, Sridharan A, Hwang M. Transtemporal brain contrast-enhanced ultrasound in children: preliminary experience in patients without neurological disorders. J Ultrasound. 2023 Mar;26(1):201-210. doi: 10.1007/s40477-022-00713-z. Epub 2022 Aug 27. PMID 36030353
- [Result] Hwang M, Tierradentro-Garcia LO, Haddad S, Poznick L, Kilbaugh T, Chiotos K. Feasibility of Contrast-Enhanced Ultrasound for Assessing Cardiac and Renal Microvascular Flow in Patients With Multisystem Inflammatory Syndrome in Children. Clin Pediatr (Phila). 2022 Mar;61(3):241-247. doi: 10.1177/00099228211073288. Epub 2022 Jan 26. No abstract available. PMID 35081803
- See also: Latest updates on COVID-19 from the European Centre for Disease Prevention and Control — https://doi.org/10.2807/1560-7917.ES.2020.25.6.2002131
- See also: Diagnosis of Acute Respiratory Syndrome Coronavirus 2 Infection by Detection of Nucleocapsid Protein — https://doi.org/10.1101/2020.03.07.20032524

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: Subjects with confirmed or probable COVID-19 will undergo CEUS of heart, kidneys and/or brain.
  Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection (if there are two injections of contrast) of the contrast agent.
  Sulfur hexafluoride lipid-type A microspheres: Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed to evaluate for dynamic bowel perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.
Period: Overall Study
Arm/Group | Study Population
Started | 4
Completed (4 patients were enrolled.) | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: Contrast-enhanced ultrasound scan with a duration of approximately 15 minutes will be performed when a COVID-19 diagnosis has been made (or is highly suspected) according to established clinical procedures. One CEUS will be performed per patient, with up to 2 intravenous injections of the contrast agent. The dosing plan will be weight-adjusted, based on a dose of 0.03 mL/kg (with a maximum dose of 2.4 mL per injection). Organ perfusion will be evaluated in the heart, kidneys, and/or brain. Clinical outcomes during hospital stay will be collected for correlation to CEUS-based measures.
Arm/Group | Study Population
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
Hospital stay [Median (Inter-Quartile Range); unit: Days] — Median hospital stay.
  Days | 7 [4 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Proportion of Patients With Normal Perfusion Versus Area(s) of Hypoperfusion in Heart, Kidneys and/or Brain
Description: Assess microvascular perfusion of the heart, kidneys and/or brain using CEUS in patients with confirmed or probable diagnosis of COVID-19.
  A sufficient diagnostic quality to analyze the ultrasound examination was accomplished in three out of four patients.
Time Frame: 15 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 3
Participants
  No microvascular perfusion defect observed | 2
  Microvascular perfusion defect observed (Left ventricular wall and kidney) | 1

ADVERSE EVENTS:
Time Frame: 15 minutes.
Arm/Group | Contrast-enhanced Ultrasonography
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Since this is an exploratory study with limited sample size, no absolute conclusions related to true microvascular impairment in MIS-C can be drawn. Whether heterogeneous results are due to the small sample, the timing of CEUS with regard to disease evolution and treatment, the use of concomitant medications, such as furosemide, a milder course of the disease, or the differing pathophysiology between MIS-C and primary COVID-19 infection in adults requires additional exploration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04640038/Prot_SAP_000.pdf